CLINICAL TRIAL: NCT05042882
Title: Early Enteral vs. Oral Nutrition After Whipple Procedure: a Multicentric Randomized Controlled Trial
Brief Title: Enteral vs. Oral Nutrition After Pancreatoduodenectomy
Acronym: NUTRIWHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Gaëtan-Romain Joliat, Principal Investigator, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-00724
Record Dates: First submitted 2021-08-30; First posted 2021-09-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pancreaticoduodenectomy; Malnutrition; Postoperative Complications
Keywords: Enteral nutrition; Oral nutrition; Pancreatoduodenectomy; Whipple operation; Pancreas surgery; Morbidity
MeSH Terms: conditions — Malnutrition; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early enteral nutrition (Experimental): Intervention group: enteral nutrition from the first postoperative night until 50% of caloric requirements are covered by oral nutrition. Enteral nutrition will start at a flow of 250 ml/12h. If tolerated, enteral nutrition will be increased to 500 ml/12h on postoperative day 1, 750 ml/12h on postoperative day 2, and 1000 ml/12h on postoperative day 3. A hypercaloric enteral nutrition will be used (Isosource Energy Fibre or similar).
  Interventions: Dietary Supplement: Early enteral nutrition
- Oral nutrition (No Intervention): Control group: patients will receive standardized oral nutrition. The night after the operation, patients will be allowed to have free drinks. On postoperative day 1, they will receive bouillons, creams, yogurts, and drinks >2 l. On postoperative day 2, they will receive a light diet. On postoperative day 3, they will receive half portion of normal diet and on postoperative day 4 normal diet.

INTERVENTIONS:
Dietary Supplement: Early enteral nutrition — Enteral nutrition via nasojejunal tube
  Arms: Early enteral nutrition

SUMMARY:
Patients suffering from pancreas cancer as well as patients with chronic pancreatitis or requiring pancreas surgery often are in a compromised nutritional status. Nutritional support should therefore be started early during the postoperative course to prevent further malnutrition, as it is an important risk factor to develop complications. Recently, several studies have shown that early enteral nutrition (EEN) could shorten length of stay, reduce postoperative infections and mortality, and decrease costs when compared with total parenteral nutrition (TPN) in gastrointestinal cancer surgery. After pancreatoduodenectomy (PD), EEN has been shown to reduce early and late complications, infections, and readmission rates. It is nevertheless currently not clear if EEN improves the short-term outcomes after PD compared to oral nutrition.

The primary objective of the study is to assess the impact of EEN on postoperative morbidity after PD, according to the Comprehensive Complication Index. Secondary objectives are to assess the impact of EEN on major postoperative complications, according to Clavien classification, specific complications, length of stay, readmission rates, quality of life, metabolic stress and nutritional response after PD.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for elective open pancreatoduodenectomy.
* Patient ≥18 years old.
* Patient at nutritional risk, i.e., with Nutrition Risk Screening (NRS) ≥3.
* Signed informed consent.

Exclusion Criteria:

* Patient not able to give informed consent as documented by signature of consent form (e.g., vulnerable patients).
* Enteral feeding already initiated preoperatively.
* Language barrier.
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders (i.e., eating disorders and bipolar disorders), or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication Index | Postoperative day 90
  Index measuring all complications for a patient

SECONDARY OUTCOMES:
Severe postoperative complications | Postoperative day 90
  Dindo-Clavien >II
Specific complications after pancreatoduodenectomy | Postoperative day 90
  SSI, DGE, POPF, PPH, biliary fistula, gastrojejunal anastomosis fistula, pancreatitis
Length of stay | Up to 90 days
  From operation day to hospital discharge
Readmission | Postoperative day 90
  Hospital readmission due to surgical complications
Patients' quality of life | Preoperatively and at 30 and 90 days after the operation
  EORTC questionnaires
Metabolic response to enteral nutrition | Preoperatively and twice weekly during the first postoperative week
  Laboratory results
Body composition | Preoperatively and on the day when patients leave the hospital after the operation
  Bioelectrical impedance analysis
Muscular measure | Preoperatively and on the day when patients leave the hospital after the operation
  Handgrip strength measure
Resting energy expenditure | On postoperative day 5
  Indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan-Romain Joliat, MD, Principal Investigator — University of Lausanne Hospitals; Markus Schäfer, MD, Study Director — University of Lausanne Hospitals; Nicolas Demartines, MD, Study Chair — University of Lausanne Hospitals
Locations (3):
- Hôpital Cochin-Port Royal, AP-HP, Paris, France
- Switzerland (2):
  - Lausanne University Hospital (CHUV), Lausanne, Canton of Vaud
  - Regional Hospital of Lugano, Lugano, Canton Ticino

REFERENCES:
- [Derived] Joliat GR, Martin D, Labgaa I, Melloul E, Uldry E, Halkic N, Fotsing G, Cristaudi A, Majno-Hurst P, Vrochides D, Demartines N, Schafer M. Early enteral vs. oral nutrition after Whipple procedure: Study protocol for a multicentric randomized controlled trial (NUTRIWHI trial). Front Oncol. 2022 Jun 28;12:855784. doi: 10.3389/fonc.2022.855784. eCollection 2022. PMID 35865476